CLINICAL TRIAL: NCT03714113
Title: Clinical Significance of Donor-specific Anti-HLA Antibodies Monitoring in Kidney Transplant Recipients
Brief Title: Donor-specific Anti-HLA Antibodies Monitoring in Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DI2017 002147
Record Dates: First submitted 2018-10-03; First posted 2018-10-22 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Kidney Transplant Rejection
Keywords: Donor-specific antibodies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kidney transplant recipients. (Experimental): Patients who undergo kidney transplant in 2018 or 2019.
  Interventions: Diagnostic Test: Anti-HLA donor-specific antibodies monitoring

INTERVENTIONS:
Diagnostic Test: Anti-HLA donor-specific antibodies monitoring — Monitoring anti-HLA donor-specific antibodies in the patients serum at the time of kidney transplantation and 3, 12 and 24 months after the procedure. Blood samples from patients will be collected.

SUMMARY:
The aim of this study is to evaluate whether anti-HLA donor-specific antibodies monitoring can be used as an effective tool for stratification of immunological risk in Polish kidney transplant recipients.

DETAILED DESCRIPTION:
Monitoring of immune response is one of the most important goals in the management of the patients after kidney transplantation. Researchers and clinicians are trying to extend the survival of the renal graft. Currently, it is believed that the main cause of late transplant loss is antibody-mediated rejection (ABMR). Anti-HLA donor-specific antibodies (DSA) are a proven risk factor for the development of humoral rejection and transplant loss. Antibodies in sensitized recipients occur before transplantation (preformed) or may develop de novo (in 13% -30% of patients).

DSA damage the graft in various mechanisms (complement activation, direct influence on endothelial cells, antibody-dependent cytotoxicity) leading to different clinical-morphological phenotypes. The pathogenicity of DSA is determined by number of their additional characteristics, such as: class, specificity, strength, C1q complement binding, IgG subclass . Monitoring the presence of DSA in the kidney recipient serum with the determination of their characteristics may improve the stratification of the risk of immunological loss of the renal allograft.

There is no effective treatment for ABMR, hence DSA monitoring allows for early intervention such as biopsy or modification of immunosuppressive therapy at an early stage of rejection.

ELIGIBILITY:
Inclusion Criteria:

* Deceased-donor kidney transplant recipient
* Older than 18 years
* Written consent by the patient

Exclusion Criteria:

* Younger than 18 years
* Lack of written consent by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Presence of anti-HLA donor-specific antibodies. | 24 months
  Binary variable (positive/negative).

SECONDARY OUTCOMES:
Mean fluorescence intensity (MFI) of anti-HLA DSA. | 24 months
  Assessed when anti-HLA DSA positive. Mean fluorescence intensity (MFI) of anti-HLA DSA. [units]
Presence of C1q complement binding anti-HLA DSA. | 24 months
  Assessed when anti-HLA DSA positive. Binary variable (positive/negative).
Presence of IgG1 subclass of anti-HLA DSA. | 24 months
  Assessed when anti-HLA DSA positive. Binary variable (positive/negative).
Presence of IgG2 subclass of anti-HLA DSA. | 24 months
  Assessed when anti-HLA DSA positive. Binary variable (positive/negative).
Presence of IgG3 subclass of anti-HLA DSA. | 24 months
  Assessed when anti-HLA DSA positive. Binary variable (positive/negative).
Presence of IgG4 subclass of anti-HLA DSA. | 24 months
  Assessed when anti-HLA DSA positive. Binary variable (positive/negative).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Transplantation Medicine, Nephrology and Internal Medicine, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided